CLINICAL TRIAL: NCT01996254
Title: A Randomized, Double-Blinded, Placebo-Controlled, Multicenter Pilot Study of the SPRINT Peripheral Nerve Stimulation (PNS) System for the Treatment of Post-Amputation Pain
Brief Title: Electrical Stimulation for the Treatment of Post-Amputation Pain Using the SPRINT System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPR Therapeutics, Inc. (Industry)
Collaborators: NDI Medical, LLC (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0123-CSP-000
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Post-Amputation Pain; Phantom Limb Pain; Residual Limb Pain
Keywords: electrical stimulation; neurostimulation; neuromodulation; post-amputation pain; phantom limb pain; residual limb pain; neuropathic pain; amputee pain
MeSH Terms: conditions — Phantom Limb; Neuralgia | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPRINT Group 1 (Experimental): Subjects in Group 1 will have a Lead placed in the residual limb in the upper leg. These subjects will then use the SPRINT Peripheral Nerve Stimulation (PNS) System and will receive electrical stimulation for 8 weeks.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System
- SPRINT Group 2 (Sham Comparator): Subjects in Group 2 will have a Lead placed in the residual limb in the upper leg. These subjects will then use the SPRINT Peripheral Nerve Stimulation (PNS) System for a total of 8 weeks. They will receive 4 weeks of stimulation and 4 weeks with no stimulation.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System

INTERVENTIONS:
Device: SPRINT Peripheral Nerve Stimulation (PNS) System — The SPRINT System is an Investigational Device which delivers mild electrical stimulation to nerves in the residual limb. The SPRINT System includes a small wire (called a "Lead") that is placed through the skin in the upper leg. It also includes a device worn on the body that delivers stimulation (called the SPRINT Stimulator).
  Other Names: SPRINT System, SPRINT; Smartpatch System, Smartpatch

SUMMARY:
The purpose of this study is to determine if electrical stimulation (small levels of electricity) can safely and effectively reduce post-amputation pain. This study involves a device called the SPRINT System. The SPRINT System delivers mild electrical stimulation to nerves in the residual limb. The SPRINT System includes a small wire (called a "lead") that is placed through the skin in the upper leg. It also includes a device worn on the body that delivers stimulation (called the SPRINT Stimulator).

ELIGIBILITY:
Key Inclusion Criteria:

* At least 18 years old
* Traumatic lower extremity amputation(s)
* Healed amputation and healthy residual limb based upon the investigator's evaluation

Key Exclusion Criteria:

* Change of prescribed medications affecting pain within the past 4 weeks
* Compromised immune system based on medical history
* Implanted electronic device
* Bleeding disorder
* History of valvular heart disease
* Confounding central nervous system injuries and disorders
* History of recurrent skin infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Boggs, PhD, Principal Investigator — SPR Therapeutics, Inc.
Locations (10):
- United States (10):
  - Arizona Pain, Scottsdale, Arizona
  - University of California San Diego, La Jolla, California
  - Denver Clinic for Extremities at Risk, Denver, Colorado
  - International Spine, Pain and Performance Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Northwestern University, Chicago, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Ainsworth Institute of Pain Management, New York, New York
  - Center for Clinical Research, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Gilmore CA, Ilfeld BM, Rosenow JM, Li S, Desai MJ, Hunter CW, Rauck RL, Nader A, Mak J, Cohen SP, Crosby ND, Boggs JW. Percutaneous 60-day peripheral nerve stimulation implant provides sustained relief of chronic pain following amputation: 12-month follow-up of a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2019 Nov 17:rapm-2019-100937. doi: 10.1136/rapm-2019-100937. Online ahead of print. PMID 31740443
- [Derived] Gilmore C, Ilfeld B, Rosenow J, Li S, Desai M, Hunter C, Rauck R, Kapural L, Nader A, Mak J, Cohen S, Crosby N, Boggs J. Percutaneous peripheral nerve stimulation for the treatment of chronic neuropathic postamputation pain: a multicenter, randomized, placebo-controlled trial. Reg Anesth Pain Med. 2019 Jun;44(6):637-645. doi: 10.1136/rapm-2018-100109. Epub 2019 Apr 5. PMID 30954936
- See also: Sponsor's Website — http://www.sprtherapeutics.com
- See also: Collaborator's Website — http://www.ndimedical.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in 10-2013 (with the first subject enrolling 12-2013) and was concluded in 05-2018. Subjects were screened from a pool of candidates experiencing chronic post-amputation pain.
Pre-assignment Details: Participants in the Initial Study Design Arm were only assessed for Safety (Adverse Events).
Groups:
- Initial Study Design Subjects: Subjects who were consented and enrolled under the initial design of the study. These subjects are included in the Safety Set.
- Group 1 (Treatment Group, Revised Study Design): Treatment Group subjects were consented and enrolled under the revised study design. These subjects had at least one Lead placed and received electrical stimulation therapy.
- Group 2 (Control Group, Revised Study Design): Control Group subjects were consented and enrolled under the revised study design. These subjects had at least one Lead placed and received sham stimulation therapy.
Period: Overall Study
Arm/Group | Initial Study Design Subjects | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Started | 5 | 14 | 14
Safety Set (All subjects that underwent Lead placement) | 5 | 14 | 14
Full Analysis Set (Subjects from the Revised Study Design that enrolled and met all eligibility prior to Lead placement) | 0 | 12 | 14
Long Term Analysis Set (Full Analysis Set with imputed data for missed visits and exclusion due to early termination.) | 0 | 12 | 14
Per Protocol Set (Full Analysis Set with adequate diary completion, paresthesia coverage, and continued eligibility) | 0 | 10 | 13
Completed | 4 | 9 | 6
Not Completed | 1 | 5 | 8
Not completed — Change in Eligibility | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 4
Not completed — Lost to Follow-up | 1 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: Subjects who were consented, randomized, and met all eligibility criteria prior to Lead placement
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design) | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (12.3) | 45.0 (13.2) | 46.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 14 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Median (Full Range); unit: kg per square meter] — Population: Height was not collected for 1 of the 12 (Group 1) participants so BMI was not able to be calculated for that participant. This accounts for the difference in number analyzed in this row from the 26 overall.
  kg per square meter
    number analyzed (Participants) | 11 | 14 | 25
    (all) | 26.5 [15.6 to 43.6] | 30.8 [23.0 to 34.6] | 27.4 [15.6 to 43.6]
Time Since Amputation [Median (Full Range); unit: Years] | 5.7 [0.3 to 16.4] | 4.8 [0.4 to 31.1] | 5.0 [0.3 to 31.1]
Baseline Beck Depression Inventory Score [Median (Full Range); unit: units on a scale] — The Beck Depression Inventory (BDI), version II is a survey used to measure depression severity. Scores from 0-13 indicate minimal depression, 14-19 mild depression, 20-28 moderate depression, and 29-63 severe depression. The score range is 0 to 63.
  units on a scale | 6.5 [0.0 to 20.0] | 12.5 [4.0 to 19.0] | 11.0 [0.0 to 20.0]
Location of Amputation [Count of Participants; unit: Participants]
  Above Knee | 10 | 5 | 15
  Below Knee | 2 | 9 | 11
Side of Amputation [Count of Participants; unit: Participants]
  Left Side | 8 | 6 | 14
  Right Side | 3 | 7 | 10
  Both Sides (Bilateral) | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Group 1 (Treatment) and Group 2 (Control) Subjects That Achieved ≥ 50% Reduction in All Qualifying Areas of Pain in the First 4 Weeks of Treatment
Description: Subjects completed daily diaries to record their average daily pain intensity scores for each qualifying region of pain (phantom limb pain and/or residual limb pain). These pain intensity questions were excerpted from the Brief Pain Inventory - Short Form Question 5 (BPI-5). The BPI-5 is an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." Post-amputation pain intensity scores were determined for each subject by taking the mean of the daily average pain intensity scores from their diaries at Baseline compared to the mean score for the same region(s) of pain reported over 4 weeks after the Start of Treatment (i.e., the average of all diary scores during this period). Subjects that achieved ≥ 50% reduction in their qualifying area(s) of pain were considered successful. Missing diary data were replaced using 1-week BPI-5 recall; if recall scores were unavailable, baseline values were imputed.
Time Frame: Baseline and Weeks 1-4 Post-Start of Treatment
Population: Full Analysis Set: Subjects who were consented, randomized, and met all eligibility criteria prior to Lead placement
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 12 | 14
Participants | 7 | 2

2. Primary Outcome: Number of Subjects That Experienced at Least One Study-Related Adverse Event in Treatment and Control Groups
Description: At each study visit following the baseline assessment at Visit 1, subjects were questioned if any changes in their medical status or condition had occurred since their previous visit. If the subject experienced a change that was an adverse event, an Adverse Event Form was completed by the site. The number of subjects that experienced at least one study-related adverse event is reported here.
Time Frame: Each participant enrolled was assessed for adverse events from the time of informed consent through the 12-month follow up visit. The total assessment period was approximately 13 months for each participant.
Population: Safety Set: All subjects that underwent Lead placement.
Measure: Count of Participants; unit: Participants
Groups:
- Initial Study Design Subjects: Subjects who were consented and enrolled under the initial design of the study.
Arm/Group | Initial Study Design Subjects | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 5 | 14 | 14
Participants | 0 | 5 | 8

3. Secondary Outcome: Number of Group 1 (Treatment) Subjects That Experienced ≥ 50% Reduction in All Qualifying Areas of Pain During Weeks 5-8 Compared to Group 2 (Control) Subjects During Weeks 1-4
Description: Subjects completed daily diaries to record their average daily pain intensity scores for each qualifying region of pain (phantom limb pain and/or residual limb pain). These pain intensity questions were excerpted from the Brief Pain Inventory - Short Form Question 5 (BPI-5) on a scale from 0 to 10, where 0 indicates no pain and 10 indicates pain as bad as you can imagine. Post-amputation pain intensity scores were determined by taking the mean of the daily average pain intensity scores at baseline and over weeks 5-8 post-start of treatment for Group 1 subjects and over weeks 1-4 post-start of treatment for Group 2 subjects. Subjects that achieved ≥ 50% reduction in their qualifying area(s) of pain were considered successful. Missing diary data were replaced using the bi-weekly BPI-5 recall scores; if unavailable, the BPI-5 recall from the follow-up visit was used. The number of successes in each group is reported.
Time Frame: Baseline and Weeks 1-8 Post-Start of Treatment
Population: Full Analysis Set: Subjects from the Revised Study Design that enrolled and met all eligibility prior to Lead placement.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 12 | 14
Participants | 8 | 2

4. Secondary Outcome: Proportion of Subjects That Experienced ≥ 50% Reduction in All Qualifying Areas of Pain at Months 3-12 Post-Start of Treatment
Description: Subjects were asked to recall and rate their average pain intensity over the past week (BPI-SF question 5) for each qualifying area of pain (phantom and/or residual limb pain) on a scale from 0 to 10, where 0 indicates no pain and 10 indicates pain as bad as you can imagine. The average pain intensity score(s) at baseline were compared to the same region(s) of pain at monthly intervals from months 3-12 post-start of treatment (SOT). Subjects that achieved ≥ 50% reduction in their qualifying area(s) of pain were considered successful. Certain time points for Group 2 (i.e., after crossover) were considered exploratory, but are reported with this outcome measure for ease of data entry and readability.
Time Frame: 3-months Post-SOT, 4-months Post-SOT, 5-months Post-SOT, 6-months Post-SOT, 7-months Post-SOT, 8-months Post-SOT, 9-months Post-SOT, 10-months Post-SOT, 11-months Post-SOT, and 12-months Post-SOT
Population: Long Term Analysis Set: Subjects from the Revised Study Design that enrolled and met all eligibility prior to Lead placement with imputed data for missed visits. Covarities in the imputation model included age, gender, ethnicity, race, time since amputation, location of amputation, and baseline average pain intensity score(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 12 | 14
Participants
  3-months Post-Start of Treatment: number analyzed (Participants) | 10 | 10
  3-months Post-Start of Treatment | 5 | 0
  4-months Post-Start of Treatment: number analyzed (Participants) | 10 | 8
  4-months Post-Start of Treatment | 7 | 1
  5-months Post-Start of Treatment: number analyzed (Participants) | 10 | 7
  5-months Post-Start of Treatment | 5 | 0
  6-months Post-Start of Treatment: number analyzed (Participants) | 10 | 7
  6-months Post-Start of Treatment | 4 | 0
  7-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  7-months Post-Start of Treatment | 5 | 0
  8-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  8-months Post-Start of Treatment | 6 | 0
  9-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  9-months Post-Start of Treatment | 6 | 0
  10-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  10-months Post-Start of Treatment | 5 | 0
  11-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  11-months Post-Start of Treatment | 6 | 0
  12-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  12-months Post-Start of Treatment | 6 | 1

5. Secondary Outcome: Proportion of Subjects That Experienced ≥50% Reduction in Average Pain Interference With Daily Activities
Description: Degree of post-amputation pain that interfered with 7 aspects of daily life was rated [scale (0 to 10) with higher scores indicating greater interference]. The 7 individual scores were averaged to provide an overall pain interference score. Pain interference questions (Brief Pain Inventory - Short Form Question 9) were used for each qualifying area of pain (phantom and/or residual limb pain). Group 1 subjects: baseline average pain interference scores were compared to average pain interference scores for the same region(s) of pain at each monthly interval after the start of therapy. Group 2 subjects: baseline average pain interference scores were compared to their average score at the end of 4 weeks. Proportion of successes (subjects that experienced ≥50% reduction in average pain interference scores) is reported. Certain time points for Group 2 (i.e., after crossover) were considered exploratory but are being reported here for ease of data entry and readability.
Time Frame: Baseline, 4-weeks Post-Start of Treatment (SOT), 8-weeks Post-SOT, 3-months Post-SOT, 4-months Post-SOT, 5-months Post-SOT, 6-months Post-SOT, 7-months Post-SOT, 8-months Post-SOT, 9-months Post-SOT, 10-months Post-SOT, 11-mo Post-SOT, & 12-mo Post-SOT
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 12 | 14
Participants
  4-weeks Post-Start of Treatment: number analyzed (Participants) | 11 | 13
  4-weeks Post-Start of Treatment | 6 | 2
  8-weeks Post-Start of Treatment: number analyzed (Participants) | 11 | 11
  8-weeks Post-Start of Treatment | 9 | 2
  3-months Post-Start of Treatment: number analyzed (Participants) | 10 | 10
  3-months Post-Start of Treatment | 6 | 2
  4-months Post-Start of Treatment: number analyzed (Participants) | 10 | 8
  4-months Post-Start of Treatment | 7 | 4
  5-months Post-Start of Treatment: number analyzed (Participants) | 10 | 7
  5-months Post-Start of Treatment | 7 | 2
  6-months Post-Start of Treatment: number analyzed (Participants) | 10 | 7
  6-months Post-Start of Treatment | 5 | 2
  7-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  7-months Post-Start of Treatment | 6 | 2
  8-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  8-months Post-Start of Treatment | 5 | 0
  9-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  9-months Post-Start of Treatment | 5 | 0
  10-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  10-months Post-Start of Treatment | 5 | 2
  11-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  11-months Post-Start of Treatment | 5 | 2
  12-months Post-Start of Treatment: number analyzed (Participants) | 9 | 6
  12-months Post-Start of Treatment | 5 | 2

6. Secondary Outcome: Proportion of Group 1 (Treatment) Subjects That Experienced ≥ 10-point Reduction in Pain Disability at Monthly Intervals Post-Start of Treatment Compared to Group 2 (Control) Subjects at Week 4 Post-Start of Treatment
Description: The Pain Disability Index (PDI) is a validated survey measuring the degree pain disrupts 7 categories of life activities on a scale from 0 to 10, with higher scores indicating greater disability. The 7 scores were summed for each subject to provide an overall pain disability score. For Group 1 subjects, the baseline average PDI score was compared to PDI scores at monthly intervals. For Group 2 subjects, the baseline average PDI score was compared to their PDI score at the end of 4 weeks. The proportion of successes (subjects reporting ≥10 point reduction in PDI scores from baseline) are reported for Group 1 subjects. Certain time points for Group 2 (i.e., after crossover) were considered exploratory but are being reported within this outcome measure for ease of data entry and readability.
Time Frame: as for outcome 5
Population: Full Analysis Set: Subjects from the Revised Study Design that enrolled and met all eligibility prior to Lead placement.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 12 | 14
Participants
  4-weeks Post-Start of Treatment: number analyzed (Participants) | 10 | 13
  4-weeks Post-Start of Treatment | 6 | 10
  8-weeks Post-Start of Treatment: number analyzed (Participants) | 9 | 11
  8-weeks Post-Start of Treatment | 8 | 9
  3-months Post-Start of Treatment: number analyzed (Participants) | 9 | 10
  3-months Post-Start of Treatment | 7 | 7
  4-months Post-Start of Treatment: number analyzed (Participants) | 7 | 8
  4-months Post-Start of Treatment | 6 | 7
  5-months Post-Start of Treatment: number analyzed (Participants) | 9 | 7
  5-months Post-Start of Treatment | 7 | 6
  6-months Post-Start of Treatment: number analyzed (Participants) | 7 | 7
  6-months Post-Start of Treatment | 5 | 4
  7-months Post-Start of Treatment: number analyzed (Participants) | 8 | 6
  7-months Post-Start of Treatment | 6 | 4
  8-months Post-Start of Treatment: number analyzed (Participants) | 8 | 5
  8-months Post-Start of Treatment | 6 | 4
  9-months Post-Start of Treatment: number analyzed (Participants) | 8 | 4
  9-months Post-Start of Treatment | 5 | 4
  10-months Post-Start of Treatment: number analyzed (Participants) | 6 | 4
  10-months Post-Start of Treatment | 5 | 4
  11-months Post-Start of Treatment: number analyzed (Participants) | 6 | 4
  11-months Post-Start of Treatment | 5 | 4
  12-months Post-Start of Treatment: number analyzed (Participants) | 7 | 4
  12-months Post-Start of Treatment | 5 | 3

7. Secondary Outcome: Depression at Monthly Intervals After Start of Therapy
Description: The Beck Depression Inventory (BDI-II) is a validated, 21-question survey used to measure depression severity. Question are rated on a scale from 0 to 3, and the scores from each question are totaled to provide an overall score ranging between 0 to 63. Scores from 0-13 indicate minimal depression, 14-19 mild depression, 20-28 moderate depression, and 29-63 severe depression. Group 1 subjects: baseline BDI-II score was compared to BDI-II scores at monthly intervals. Group 2 subjects: baseline BDI-II score was compared to their BDI-II score at the end of 4 weeks. The percent change from baseline to each monthly interval is reported. Certain timepoints for Group 2 (i.e., after crossover) were considered exploratory but are being reported within this outcome measure for ease of data entry and readability.
Time Frame: as for outcome 5
Population: Full Analysis Set: Subjects from the Revised Study Design that enrolled and met all eligibility prior to Lead placement.
Measure: Median (Full Range); unit: percent change
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 12 | 14
percent change
  4-weeks Post-Start of Treatment: number analyzed (Participants) | 10 | 13
  4-weeks Post-Start of Treatment | -17.69 [-100.00 to 50.00] | -11.76 [-91.67 to 136.36]
  8-weeks Post-Start of Treatment: number analyzed (Participants) | 9 | 11
  8-weeks Post-Start of Treatment | -50.00 [-100.00 to 100.00] | -15.38 [-100.00 to 129.41]
  3-months Post-Start of Treatment: number analyzed (Participants) | 9 | 10
  3-months Post-Start of Treatment | -55.00 [-100.00 to 177.78] | -10.00 [-50.00 to 154.55]
  4-months Post-Start of Treatment: number analyzed (Participants) | 7 | 8
  4-months Post-Start of Treatment | -75.00 [-100.00 to 111.11] | -35.29 [-70.59 to 70.59]
  5-months Post-Start of Treatment: number analyzed (Participants) | 9 | 7
  5-months Post-Start of Treatment | -75.00 [-100.00 to 88.89] | -47.06 [-100.00 to 70.59]
  6-months Post-Start of Treatment: number analyzed (Participants) | 7 | 7
  6-months Post-Start of Treatment | -50.00 [-100.00 to 22.22] | 22.22 [-75.00 to 136.36]
  7-months Post-Start of Treatment: number analyzed (Participants) | 8 | 6
  7-months Post-Start of Treatment | -30.00 [-100.00 to 50.00] | 11.76 [-75.00 to 122.22]
  8-months Post-Start of Treatment: number analyzed (Participants) | 8 | 5
  8-months Post-Start of Treatment | -70.00 [-100.00 to 50.00] | -41.18 [-50.00 to 90.91]
  9-months Post-Start of Treatment: number analyzed (Participants) | 8 | 4
  9-months Post-Start of Treatment | -68.75 [-100.00 to 50.00] | -17.65 [-50.00 to 90.91]
  10-months Post-Start of Treatment: number analyzed (Participants) | 7 | 4
  10-months Post-Start of Treatment | -65.00 [-100.00 to 25.00] | -67.65 [-75.00 to 90.91]
  11-months Post-Start of Treatment: number analyzed (Participants) | 7 | 4
  11-months Post-Start of Treatment | -80.00 [-100.00 to 25.00] | -69.85 [-100.00 to 90.91]
  12-months Post-Start of Treatment: number analyzed (Participants) | 7 | 4
  12-months Post-Start of Treatment | 0.00 [-100.00 to 66.67] | -72.79 [-100.00 to 209.09]

8. Secondary Outcome: Change in Opioid Analgesic Usage From Baseline
Description: Changes in opioid analgesic usage were calculated using morphine equivalent dosing (MED) for subjects who were using opioid analgesics at baseline. Subjects completed daily diaries in which they tracked their use of analgesic medications. For Group 1 subjects, the mean daily MED from the baseline diary was compared to the mean daily MED during week 4 and week 8. For Group 2 subjects, the daily MED from the baseline diary was compared to the daily MED during week 4 only. The median percent change from baseline is reported. Certain time points for Group 2 (i.e., after crossover) were considered exploratory but are being reported within this outcome measure for ease of data entry and readability.
Time Frame: Baseline, 4-weeks Post-Start of Treatment (SOT), and 8-weeks Post-SOT
Population: Full Analysis Set: Subjects from the Revised Study Design that enrolled and met all eligibility prior to Lead placement. Only the 9 subjects that were using opioid analgesics at baseline were included in the analysis.
Measure: Median (Full Range); unit: percent change
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 12 | 14
percent change
  4-Weeks Post-Start of Treatment: number analyzed (Participants) | 4 | 5
  4-Weeks Post-Start of Treatment | 32.68 [26.32 to 100.00] | 47.17 [-55.60 to 100.00]
  8-Weeks Post-Start of Treatment: number analyzed (Participants) | 4 | 5
  8-Weeks Post-Start of Treatment | 78.79 [26.32 to 100.00] | 45.28 [-55.60 to 100.00]

9. Secondary Outcome: Percent Change in Hours of Daily Prosthetic Usage
Description: Subjects completed daily diaries in which they tracked the number of hours of their prosthetic usage. The 7-day mean prosthetic use was calculated for each subject from their baseline diary and compared to the 7-day mean from week 4 and week 8. The percent change from baseline was then calculated for each subject at each time point (i.e., 4-week median vs. baseline median and 8-week median vs. baseline median). A positive value indicates an increase in prosthetic usage.
Time Frame: Baseline, 4-weeks Post-Start of Treatment (SOT), and 8-weeks Post-SOT
Population: Full Analysis Set: Subjects from the Revised Study Design that enrolled and met all eligibility prior to Lead placement.
Measure: Median (Full Range); unit: percent change
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 12 | 14
percent change
  4-weeks Post-Start of Treatment: number analyzed (Participants) | 6 | 10
  4-weeks Post-Start of Treatment | 2.49 [-19.10 to 28.89] | 4.51 [-20.00 to 95.52]
  8-weeks Post-Start of Treatment: number analyzed (Participants) | 5 | 9
  8-weeks Post-Start of Treatment | 3.23 [-5.75 to 20.00] | 9.14 [-19.11 to 82.84]

10. Secondary Outcome: Subject Satisfaction Survey
Description: Subjects completed a sponsor-developed survey with questions pertaining to their feelings about therapy as delivered by the SPRINT Beta Stimulation System as a method for managing chronic post-amputation pain. Subjects were asked to report on their experience using the therapy. Depending on the question, subjects were asked to indicate their agreement with the question (strongly disagree, agree, neutral, disagree, strongly disagree), their comfort with the therapy (very uncomfortable, a little bit uncomfortable, fairly comfortable, very comfortable), or when pain relief was felt (immediately, a few minutes later, a few hours later, more than a day later or never). Responses are presented for key groups of questions related to the therapy whereby answer options are considered affirmative for strongly agree/agree, very easy/easy, very comfortable/comfortable.
Time Frame: Visit 11 (8-weeks post-Start of Treatment (SOT))
Population: Of the 28 total subjects, 14 subjects that used one version of the stimulator (Sprint Beta) were asked to complete subject surveys and 6 of the 14 responded. Results are presented for the 6 surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
Number analyzed (Participants) | 3 | 3
Participants
  Pain relief (w/stim) immediate/within a few hours | 3 | 3
  Stimulation felt comfortable/soothing/tolerable | 3 | 3
  Prefer stimulation to pain medications | 3 | 3
  Would recommend therapy | 3 | 2
  Tolerated lead placement w/some or no discomfort | 3 | 3
  Would like to have used stimulation longer | 3 | 2

ADVERSE EVENTS:
Time Frame: Each participant enrolled was assessed for adverse events from the time of informed consent through the 12-month follow up visit. The total assessment period was approximately 13 months for each participant.
Arm/Group | Initial Study Design Subjects | Group 1 (Treatment Group, Revised Study Design) | Group 2 (Control Group, Revised Study Design)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/14 | 1/14
Other Adverse Events (participants affected / at risk) | 0/5 | 8/14 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Study Design Subjects (N=5) | Group 1 (Treatment Group, Revised Study Design) (N=14) | Group 2 (Control Group, Revised Study Design) (N=14)
Car accident (Social circumstances) | 1 (1) | 0 (0) | 0 (0) — Not study-related
Patellar Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Not study-related
Gallstones (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Not study-related
Leg Pain/Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Not study-related
Pleuritic Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Not study-related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Study Design Subjects (N=5) | Group 1 (Treatment Group, Revised Study Design) (N=14) | Group 2 (Control Group, Revised Study Design) (N=14)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — Not study related
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Not study related
Tiredness/Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0) — One event was study related, and the other was not
Cold/Flu/Sinus infection (General disorders) | 0 (0) | 1 (1) | 1 (1) — Not study related
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) — Unable to determine relationship
Broken bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related
Pain and tenderness from procedure (Product Issues) | 0 (0) | 0 (0) | 3 (3) — Study related
Unpleasant painful stimulation (Product Issues) | 0 (0) | 2 (2) | 0 (0) — Study related
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Not study related
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) — Not study related
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) — Not study related
Itching irritation or bruising from SPRINT pads (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) — Study related
Skin irritation/redness at Lead exit site (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (3) — Study related
Itching or irritation from bandages and/or belt (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (4) — Study related
Non-specified skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — One event was study related, and the other was not
Blister/abcess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — Not study related
Surgery (Surgical and medical procedures) | 0 (0) | 1 (2) | 1 (1) — Not study related
Fall (Social circumstances) | 0 (0) | 1 (1) | 1 (1) — Not study related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT01996254/Prot_SAP_000.pdf